CLINICAL TRIAL: NCT04581967
Title: Pharmacogenetic Risk Factors of Doxorubicin-Cyclophosphamide Chemotherapy Related Toxicities in Breast Cancer Patients
Brief Title: Study of CYP2C19 and ALDH3A1 Polymorphisms in Breast Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Damanhour University (Other)
Collaborators: Al-Azhar University (Other); National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Amira Bisher,PhD, principal investigator, Damanhour University
Other Study IDs: 201819010.4
Record Dates: First submitted 2020-04-22; First posted 2020-10-09 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2020-08

CONDITIONS: Breast Cancer Patients
MeSH Terms: interventions — Amplified Fragment Length Polymorphism Analysis; Polymorphism, Single Nucleotide; Neoadjuvant Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA extract by extraction kits from whole blood
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Genetic: polymorphism analysis — * DNA will be purified from whole blood samples by commercial DNA isolation kits.
  * Genotyping and genetic polymorphism detection for some metabolic enzymes genes will be performed by real time PCR.
  Other Names: single nucleotide polymorphism
Drug: Doxorubicin-Cyclophosphamide regimen — Treatment with a combination of Doxorubicin and Cyclophosphamide, This regimen comprises 60 mg/m² Doxorubicin and 600 mg/m² Cyclophosphamide administered intravenously on day 1 of each 21-day cycle, and repeated for a total of four cycles.
  Other Names: chemotherapy treatment

SUMMARY:
Genetic polymorphisms of metabolic enzymes may influence the metabolism of Doxorubicin-Cyclophosphamide regimen in breast cancer patients.

the investigators want to

1. evaluate the frequency or incidence of the genetic polymorphisms of CYP2C19 and ALDH3A1 in breast cancer patients, and
2. analyze the association between the genetic polymorphisms of CYP2C19 and ALDH3A1 and toxicities in breast cancer patients treated by Doxorubicin-Cyclophosphamide regimen therapy.

DETAILED DESCRIPTION:
Breast cancer refers to the erratic growth and proliferation of cells that originate in the breast tissue, most commonly from the inner lining of milk ducts (ductal cancers) or the lobules that supply the ducts with milk (lobular cancers). Breast cancer is about 100 times more common in women than in men, although males tend to have poorer outcomes due to delays in diagnosis. Alteration in hormonal level and Family history of breast cancer are risk factors for breast cancer.

The classic symptom for breast cancer is a lump found in the breast or armpit. Doing monthly breast self-exam (BSE) is a great way to be familiar with the breasts' texture, cyclical changes, size, and skin condition. Breast cancer is usually diagnosed by biopsy of nodule detected by mammogram or by palpitation.

Today there are so many approaches, which can be made for the treatment of breast cancer such as surgery, radiation therapy, chemotherapy, hormonal therapy and recently nanotechnology and gene therapy. Chemotherapy is the use of anti-cancer drugs to treat cancerous cells. The differences in patients' response to the same medication, toxicity included, are one of the major problems in breast cancer treatment.

Chemotherapy toxicity makes a significant clinical problem due to decreased quality of life, prolongation of treatment and reinforcement of negative emotions associated with therapy. Four cycles of doxorubicin and cyclophosphamide (AC) chemotherapy regimen has become a standard regimen. No chemotherapy regimen administered for four cycles has proven to be superior to AC. The undeniable advantage of this therapy scheme is low cost of treatment, its proven efficacy and mostly acceptable toxicity. Hematological (neutropenia and anemia) and gastrointestinal (nausea, vomiting and mucositis) toxicities are common in patients treated with AC regimen.

Doxorubicin is metabolized by the CBR (carbonyl reductase) enzymes to its active component. Similarly cyclophosphamide, the cell cycle nonspecific prodrug, requires activation by a number of different cytochrome P450 enzymes, mainly of CYP2C family. The transport systems are also crucial for the treatment outcome, as both importers and exporters are responsible for the cellular drugs' concentration. It is expected that any variation that affects metabolic enzymes and transporter activity would be reflected in not only the response to treatment, but also in the development of drug-related toxicity. Each of these enzymes and transporter genes is known to exhibit a degree of genetic variation, characterized by single nucleotide polymorphisms (SNPs). In particular, there have been few investigations of the possible influence of variations in the genes encoding transporters and drug metabolizing enzymes relevant for the two drugs.

Pharmacogenomic analysis offers the promise that personalized regimens may be identified for individuals who might have more favorable outcomes with certain chemotherapies. Specifically, because genetic variation in metabolic enzymes is one determinant of drug concentration, pharmacogenomics has been proposed as an approach to tailor drug choice or dose to optimize efficacy and reduce toxicity of cancer treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of breast cancer.
2. Age ranging from 18 to 75 years old female.
3. Patients will take Doxorubicin-Cyclophosphamide regimen as chemotherapy treatment.

Exclusion Criteria:

1. Any other malignancy.
2. Previous treatment for metastatic disease.
3. Pregnancy or breastfeeding female.
4. Inadequate bone marrow and cardiac function.
5. Serious or uncontrolled medical conditions.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all breast cancer patients receiving either adjuvant or neoadjuvant therapy in National Cancer Institute
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-10-15 (Estimated); Primary Completion 2020-12-15 (Estimated); Study Completion 2021-01-15 (Estimated)

PRIMARY OUTCOMES:
The frequency of the genetic polymorphisms of CYP2C19 in breast cancer patients | Up to 24 weeks
  the blood samples will be DNA extracted using DNA extraction kit then single nucleotide polymorphisms of CYP2C19 gene will be detected by real time PCR
The frequency of the genetic polymorphisms of ALDH3A1 in breast cancer patients | Up to 24 weeks
  the blood samples will be DNA extracted by DNA extraction kit then single nucleotide polymorphisms of ALDH3A1 gene will be detected by real time PCR

SECONDARY OUTCOMES:
Correlation between genetic polymorphisms of CYP2C19 and toxicities from Doxorubicin-Cyclophosphamide regimen therapy | up to 24 weeks
  the blood samples will be DNA extracted using DNA extraction kit then single nucleotide polymorphisms of CYP2C19 gene will be detected by real time PCR
Correlation between genetic polymorphisms of ALDH3A1 and toxicities from Doxorubicin-Cyclophosphamide regimen therapy | up to 24 weeks
  the blood samples will be DNA extracted by DNA extraction kit then single nucleotide polymorphisms of ALDH3A1 gene will be detected by real time PCR

CONTACTS AND LOCATIONS:
Overall Officials: Hoda Salem, Ass. Prof, Study Director — faculty of pharmacy, Al-Azhar university; Marwa Nabeel, Ass. Prof, Study Chair — National Cancer Institute-Cairo University; Amira Bisheer, PhD, Principal Investigator — faculty of pharmacy, Damanhour University; Esraa Khaled, B. Pharm, Principal Investigator — faculty of pharmacy, Al-Azhar University
Locations (1):
- National Cancer Institute, Cairo, Egypt

REFERENCES:
- [Background] Sharma GN, Dave R, Sanadya J, Sharma P, Sharma KK. Various types and management of breast cancer: an overview. J Adv Pharm Technol Res. 2010 Apr;1(2):109-26. PMID 22247839
- [Background] Tecza K, Pamula-Pilat J, Lanuszewska J, Butkiewicz D, Grzybowska E. Pharmacogenetics of toxicity of 5-fluorouracil, doxorubicin and cyclophosphamide chemotherapy in breast cancer patients. Oncotarget. 2018 Jan 10;9(10):9114-9136. doi: 10.18632/oncotarget.24148. eCollection 2018 Feb 6. PMID 29507678
- [Background] Jones SE, Savin MA, Holmes FA, O'Shaughnessy JA, Blum JL, Vukelja S, McIntyre KJ, Pippen JE, Bordelon JH, Kirby R, Sandbach J, Hyman WJ, Khandelwal P, Negron AG, Richards DA, Anthony SP, Mennel RG, Boehm KA, Meyer WG, Asmar L. Phase III trial comparing doxorubicin plus cyclophosphamide with docetaxel plus cyclophosphamide as adjuvant therapy for operable breast cancer. J Clin Oncol. 2006 Dec 1;24(34):5381-7. doi: 10.1200/JCO.2006.06.5391. PMID 17135639
- [Background] Montoya JE, Luna HG, Morelos AB, Catedral MM, Lava AL, Amparo JR, Cristal-Luna GR. Association of creatinine clearance with neutropenia in breast cancer patients undergoing chemotherapy with fluorouracil, doxorubicin, and cyclophosphamide (FAC). Med J Malaysia. 2013 Apr;68(2):153-6. PMID 23629563
- [Background] Bray J, Sludden J, Griffin MJ, Cole M, Verrill M, Jamieson D, Boddy AV. Influence of pharmacogenetics on response and toxicity in breast cancer patients treated with doxorubicin and cyclophosphamide. Br J Cancer. 2010 Mar 16;102(6):1003-9. doi: 10.1038/sj.bjc.6605587. Epub 2010 Feb 23. PMID 20179710
- [Background] Zhou X, Qiao G, Wang X, Song Q, Morse MA, Hobeika A, Gwin WR, Ren J, Lyerly HK. CYP1A1 genetic polymorphism is a promising predictor to improve chemotherapy effects in patients with metastatic breast cancer treated with docetaxel plus thiotepa vs. docetaxel plus capecitabine. Cancer Chemother Pharmacol. 2018 Feb;81(2):365-372. doi: 10.1007/s00280-017-3500-9. Epub 2017 Dec 14. PMID 29242966